CLINICAL TRIAL: NCT01619982
Title: Effect of Pre-operative Prophylaxis With Vancomycin on Rate of Cefazolin Non-susceptible Gram Positive Surgical Site Infections in Cardiovascular Surgery Patients
Brief Title: Pre-operative Prophylaxis With Vancomycin and Cefazolin in Pediatric Cardiovascular Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chandra Ramamoorthy, Professor, Anesthesiology, Department of Pediatric Cardiac Anesthesia, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-11112011-8670
Record Dates: First submitted 2012-03-02; First posted 2012-06-15 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Congenital Heart Diseases; Aortic Valve Disorder
MeSH Terms: conditions — Heart Defects, Congenital; Aortic Valve Disease | interventions — Cefazolin; Weights and Measures; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin 25 mg/kg body weight and vancomycin (Active Comparator): All infants < 1 year of age with congenital heart diseases requiring cardiac surgery with cardiopulmonary bypass or any patient who requires surgery involving the aorta or the aortic valve will receive both Cefazolin and Vancomycin as preoperative prophylaxis against Surgical Site Infections. This has been recommended in recently published guidelines but not evaluated in children.
  Intervention: Cefazolin 25 mg/kg body weight and Vancomycin hydrochloride 15 mg/kg body weight
  Interventions: Drug: Cefazolin 25 mg/kg body weight and Vancomycin hydrochloride
- Cefazolin only 30mg/kg body weight (Other): All infants less than one year of age with congenital heart diseases requiring cardiac surgery with cardiopulmonary bypass or all patients who required surgery involving the aorta or the aortic valve received cefazolin 30 mg/kg body weight as preoperative prophylaxis against surgical site infections
  Interventions: Drug: Cefazolin 30 mg/kg body weight

INTERVENTIONS:
Drug: Cefazolin 25 mg/kg body weight and Vancomycin hydrochloride — Cefazolin 25 mg/kg/dose administered intravenously over 5 minutes within 60 minutes of surgical incision and then re-dosed (25 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery and Vancomycin 15 mg/kg (max 1.5 gram/dose) will be administered intravenously over 1-2 hours (after completion of cefazolin infusion) For patients younger than 1 month of age, a one-time repeat dose of 15 mg/kg can be given intraoperatively 12 hours after the beginning of the first vancomycin dose if the procedure is > 12 hours in duration. For patients equal to or older than 1 month, a one-time repeat dose of 15 mg/kg (max 1.5 grams) will be given intra-operatively 8 hours after the beginning of the first vancomycin dose if the procedure is > 8 hours in duration.
  Other Names: Cefazolin: Brand Names Ancef; Vancomycin HCL: Brand name Vancocin
  Arms: Cefazolin 25 mg/kg body weight and vancomycin
Drug: Cefazolin 30 mg/kg body weight — Intervention: Drug: Cefazolin pre-operative prophylaxis
  Other Names:
  Cefazolin: Brand Names Ancef, Kefzol
  Cefazolin 30 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (30 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
  Other Names: Cefazolin: Brand Names Ancef, Kefzol
  Arms: Cefazolin only 30mg/kg body weight

SUMMARY:
The investigators hope to learn 1) if the addition of prophylaxis with vancomycin will decrease the rate of cefazolin non-susceptible surgical site infections (SSI), in high risk population 2) to develop better understanding of vancomycin and cefazolin pharmacokinetics in children undergoing cardiopulmonary bypass (CPB) 3) to assess the barriers to vancomycin dosing peri-operatively 4) to assess side effects and risks associated with peri-operative vancomycin administration. This will allow us to improve patient care by better understanding the benefits or the risks of peri-operative vancomycin administration and potentially decrease cefazolin-resistant surgical site infections.

In addition, this study gives us the opportunity to evaluate cefazolin and vancomycin pharmacokinetics (pK) on children on CPB.

The investigators will take blood samples from 20 patients. In 10 patients the investigators will do Cefazolin pK analysis and in the other 10 the investigators will do pK Vancomycin analysis. For the remainder of 292 patients, only prospective chart review will be done to determine the incidence of SSIs.

This data will be compared with 936 controls who received only Cefazolin pre-operatively as prophylaxis for SSI's.

--------------------------------------------------------------------------------

DETAILED DESCRIPTION:
With 100% compliance with the surgical infection prevention (SIP) bundle, the risk of surgical site infections (SSIs) has decreased considerably, but is still greater than the baseline rate at the best comparison hospital (2.5%). Recent analysis of SSI's in cardiovascular surgery patients identified more than half being caused by cefazolin resistant gram positive bacteria (methicillin resistant coagulase negative staphylococci- MRSE (methicillin resistant Staphylococcus epidermidis, or methicillin resistant Staphylococcus aureus- MRSA). Cefazolin is routinely given pre-operatively as surgical prophylaxis in patients undergoing cardiovascular surgery. Vancomycin is not routinely recommended for prophylaxis due to concerns of developing vancomycin resistance, however patients with MRSE and MRSA SSIs end up needing additional surgery to remove or replace infected hardware or grafts and/or additional weeks to months of intravenous vancomycin therapy. This results in significant morbidity to the children and cost to the institution. Several published guidelines suggest the use of pre-operative prophylaxis with vancomycin (alone or in conjunction with cefazolin) in instances where patients may be at higher risk for infection with MRSE or MRSA. The purpose of this study is to determine whether the addition of vancomycin to standard pre-operative prophylaxis with cefazolin in selected high risk subjects along with the full SIP bundle will decrease the incidence of cefazolin-resistant SSI's.

ELIGIBILITY:
Inclusion Criteria:

1. Patient less than or equal to 1 year of age who is undergoing cardiovascular surgery requiring CPB or patient under 18 years of age undergoing procedures involving aortic valve or aorta
2. Patients with a positive MRSA screen or a history of MRSA infections who are undergoing any cardiac surgery

Exclusion Criteria:

1. Patients who have known hypersensitivity to vancomycin or cephalosporins
2. Patients with renal insufficiency
3. Patients who have received vancomycin or cephalosporins 48 hours prior to the day of surgery
4. Patients whose surgery is due to an infection-related diagnosis such as endocarditis
5. Patients whose parents do not wish to have them receive vancomycin prophylaxis
6. Neonates born at less than 38 weeks gestational age

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gutierrez, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Derived] Ingrande J, Gutierrez K, Lemmens HJ, Verma A, Nicolau DP, Sutherland CA, Ramamoorthy C. Pharmacokinetics of Cefazolin and Vancomycin in Infants Undergoing Open-Heart Surgery With Cardiopulmonary Bypass. Anesth Analg. 2019 May;128(5):935-943. doi: 10.1213/ANE.0000000000003876. PMID 30995208

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefazolin 25 mg/kg Body Weight and Vancomycin: Cefazolin 25 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (25 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
  Vancomycin hydrochloride: Vancomycin 15 mg/kg (max 1.5 gram/dose) will be administered intravenously over 1-2 hours (after completion of cefazolin infusion). Repeat same dose intraoperatively at 8 hours or at 12 hours if patient younger than 1 month of age.
- Cefazolin 30 mg/kg Body Weight: Cefazolin 30 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (30 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
Period: Overall Study
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30 mg/kg Body Weight
Started | 20 | 12
Completed | 20 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30 mg/kg Body Weight | Total
Number analyzed (Participants) | 20 | 12 | 32
Age, Customized [Count of Participants; unit: Participants]
  0 day to 12 months | 20 | 12 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Receive Preoperative Vancomycin and Cefazolin Who Develop a Surgical Site Infection Compared to Those Whose Received Only Cefazolin.
Description: Number of patients who receive preoperative vancomycin and cefazolin who develop a surgical site infection (SSI) compared to those whose received only cefazolin. Surveillance was done with standard procedures and definitions.
Time Frame: Patients will be monitored for superficial SSIs for 30 days from the date of surgery. Patients will be monitored for 30 days for deep SSIs if no foreign material was implanted and for 1 year if foreign material is present.
Population: Pre-operative Prophylaxis With Vancomycin and Cefazolin in Pediatric Cardiovascular Surgery Patients undergoing cardiopulmonary bypass
Measure: Number; unit: participants
Groups:
- Cefazolin 25mg/kg Body Weight and Vancomycin: Cefazolin 25 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (25 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
  Vancomycin hydrochloride: Vancomycin 15 mg/kg (max 1.5 gram/dose) will be administered intravenously over 1-2 hours (after completion of cefazolin infusion). Repeat same dose intraoperatively at 8 hours or 12 hours if patient younger than 1 month of age.
- Cefazolin 30mg/kg Body Weight: Cefazolin 30 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (30 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
Arm/Group | Cefazolin 25mg/kg Body Weight and Vancomycin | Cefazolin 30mg/kg Body Weight
Number analyzed (Participants) | 20 | 12
participants | 0 | 0

2. Secondary Outcome: Cefazolin Pharmacokinetics
Description: Cefazolin Pharmacokinetics was measured as Central Volume, Peripheral Volume (Fast), Peripheral Volume (Slow)
Time Frame: Drug levels will be sampled only during the peri-operative time period (0 to 12 hours)
Population: Cefazolin pharmacokinetics were assessed only in the Cefazolin 30 mg/kg Body Weight group
Measure: Median (95% Confidence Interval); unit: L
Groups:
- Cefazolin 25 mg/kg Body Weight and Vancomycin: Cefazolin 25 mg/kg/dose administered intravenously over 5 minutes within 60 minutes of surgical incision and then re-dosed (25 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
  Vancomycin hydrochloride: Vancomycin 15 mg/kg (max 1.5 gram/dose) will be administered intravenously over 1-2 hours (after completion of cefazolin infusion). Repeat same dose intraoperatively at 8 hours or 12 hours if patient younger than 1 month of age.
- Cefazolin 30mg/kg Body Weight: Cefazolin 30 mg/kg/dose administered intravenously over 5 minutes within 60 minutes of surgical incision and then re-dosed (30 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30mg/kg Body Weight
Number analyzed (Participants) | 0 | 10
L
  Central Volume |  | 0.547 [0.408 to 0.685]
  Peripheral Volume (Fast) |  | 0.102 [0.099 to 0.103]
  Peripheral Volume (slow) |  | 0.7 [0.69 to 0.71]

3. Secondary Outcome: Cefazolin Pharmacokinetics
Description: Measured as Elimination Clearance Inter-tissue Clearance (Fast) Inter-tissue Clearance(Slow)
Time Frame: Drug levels will be sampled only during the peri-operative time period (0 to 12 hours)
Population: Cefazolin pharmacokinetics were assessed only in the Cefazolin 30 mg/kg Body Weight group
Measure: Median (95% Confidence Interval); unit: L/min
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30mg/kg Body Weight
Number analyzed (Participants) | 0 | 10
L/min
  Elimination clearance |  | 0.00396 [0.00393 to 0.00398]
  Inter-tissue Clearance (Fast) |  | 0.1 [0.1 to 0.102]
  Inter-tissue Clearance (slow) |  | 0.0231 [0.023 to 0.0232]

4. Secondary Outcome: Vancomycin Pharmacokinetics (Plasma Concentration vs Time Curve) in Children During the Peri-operative Period in Infants Undergoing Cardiac Surgery With Cardiopulmonary Bypass (CPB)
Description: Vancomycin pharmacokinetics measured as Central Volume, Peripheral Volume (Fast), Peripheral Volume (Slow)
Time Frame: Drug levels will be sampled only during the peri-operative time period (0 to 12 hours)
Population: Vancomycin pharmacokinetics were assessed only in the Cefazolin 25 mg/kg body weight and Vancomycin arm
Measure: Median (95% Confidence Interval); unit: L
Groups:
- Cefazolin 25 mg/kg Body Weight and Vancomycin: Cefazolin 25 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (25 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
  Vancomycin hydrochloride: Vancomycin 15 mg/kg (max 1.5 gram/dose) will be administered intravenously over 1-2 hours (after completion of cefazolin infusion). Repeat same dose intraoperatively at 8 hours or 12 hours if patient younger than 1 month of age.
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30mg/kg Body Weight
Number analyzed (Participants) | 10 | 0
L
  Central Volume | 0.901 [0.79 to 1.07] |
  Peripheral Volume (Fast) | 1.02 [1.0 to 1.03] |
  Peripheral Volume (Slow) | 1.81 [1.8 to 1.83] |

5. Secondary Outcome: Vancomycin Pharmacokinetics (Plasma Concentration vs Time Curve) in Children on Cardiopulmonary Bypass (CPB)
Description: Vancomycin pharmacokinetics measured as Elimination Clearance, Inter-tissue Clearance (Fast), Inter-tissue Clearance (Slow).
Time Frame: Drug levels will be sampled only during the peri-operative time period (0 to 12 hours)
Population: Vancomycin pharmacokinetics were assessed only in the Cefazolin 25 mg/kg body weight and Vancomycin arm
Measure: Median (95% Confidence Interval); unit: L/min
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30mg/kg Body Weight
Number analyzed (Participants) | 10 | 0
L/min
  Elimination Clearance | 0.00695 [0.0067 to 0.0071] |
  Inter-tissue Clearance (Fast) | 0.0554 [0.039 to 0.067] |
  Inter-tissue Clearance (Slow) | 0.0202 [0.017 to 0.026] |

6. Secondary Outcome: Count of Participants Experiencing Adverse Events Commonly Associated With Peri-operative Vancomycin Prophylaxis
Description: Will evaluate for vancomycin associated pre or intraoperative adverse events:
  1. Hypotension requiring treatment
  2. Rash, flushing or Red Man's syndrome
  3. Other changes in vital signs (decrease in baseline 02 sat, increased heart or respiratory rate, elevated body temperature) felt to be associated with vancomycin administration
  4. An event associated with vancomycin administration which results in delay in surgery
Time Frame: Adverse events to vancomycin will be assessed on each patient in the study during the time the patient is in the operating room (0-<24 hours)
Population: Only the Cefazolin 25 mg/kg Body Weight and Vancomycin groups were assessed, the Cefazolin 30mg/kg body weight did not receive vancomycin
Measure: Count of Participants; unit: Participants
Groups:
- Cefazolin 30mg/kg Body Weight: Cefazolin pre-operative prophylaxis: Cefazolin 30 mg/kg/dose administered intravenously over 5 minutes within 60 minutes of surgical incision and then re-dosed (30mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin 30mg/kg Body Weight
Number analyzed (Participants) | 20 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: Patients will be monitored for superficial SSIs for 30 days . Patients will be monitored for 30 days for deep SSIs if no foreign material was implanted and for 1 year if foreign material is implanted from the date of surgery.
Description: Superficial SSI and adverse events related to vancomycin were assessed during the study period.
Groups:
- Cefazolin30 mg/kg Body Weight: Cefazolin 25 mg/kg/dose administered intravenously over 10 minutes within 60 minutes of surgical incision and then re-dosed (25 mg/kg: maximum 2 grams/dose) every 4 hours intra-operatively depending on the duration of surgery as per standard peri-operative prophylaxis for cardiac surgery.
Arm/Group | Cefazolin 25 mg/kg Body Weight and Vancomycin | Cefazolin30 mg/kg Body Weight
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/12
Other Adverse Events (participants affected / at risk) | 0/20 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes